CLINICAL TRIAL: NCT05248074
Title: An Open-label, Randomized, Crossover Phase 1 Clinical Trial to Evaluate the Safety, Pharmacokinetic Characteristics and the Effect of Food After Administration of ABN401 in Healthy Adult Volunteers
Brief Title: To Evaluate the Safety, Pharmacokinetic and the Effect of Food After Administration of ABN401 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abion Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABN401-002
Record Dates: First submitted 2022-01-26; First posted 2022-02-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (Other): Period 1 : Single oral administration of ABN401 800 mg (3 x 250 mg + 2 x 25 mg) after an overnight fast
  Peroid 2: Single oral administration of ABN401 800 mg (3 x 250 mg + 2 x 25 mg) in fed condition. High-fat meal (over 900 kcal)
  Interventions: Other: High-fat meal (over 900 kcal); Drug: ABN401 (investigational product)
- Fed group (Other): Peroid 1: Single oral administration of ABN401 800 mg (3 x 250 mg + 2 x 25 mg) in fed condition. High-fat meal (over 900 kcal)
  Period 2: Single oral administration of ABN401 800 mg (3 x 250 mg + 2 x 25 mg) after an overnight fast
  Interventions: Other: High-fat meal (over 900 kcal); Drug: ABN401 (investigational product)

INTERVENTIONS:
Other: High-fat meal (over 900 kcal) — High-fat meal (over 900 kcal with over 35 percent fat content of total calorie) will be provided prior to IP administration. The IP will then be administered 30 minutes after the subject begins the meal.
Drug: ABN401 (investigational product) — The investigational product, ABN401 800 mg (3 x 250 mg + 2 x 25 mg) will be administered orally with approximately 240 mL of water in fasted or fed condition in accordance with the order of IP administration in an allocated sequence.

SUMMARY:
This randomized open-label, two-way crossover study is designed to evaluate the safety and pharmacokinetic characteristics of ABN401, and the effect of high-fat meal on the pharmacokinetic profiles of ABN401 and its metabolites in healthy adult volunteers.

DETAILED DESCRIPTION:
The amount of dose for a single administration is 800 mg, which will be given as three 250 mg tablets and two 25 mg tablets.

* Fasting: Single oral administration of ABN401 800 mg (3 x 250 mg + 2 x 25 mg) after an overnight fast
* Fed: Single oral administration of ABN401 800 mg (3 x 250 mg + 2 x 25 mg) in fed condition. High-fat meal (over 900kcal with over 35 percent fat content of total calorie) will be provided prior to IP administration. The IP will then be administered 30 minutes after the subject begins the meal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged over 19 years (inclusive) at the time of screening
2. Subjects weighing at least 50.0 kg with a BMI between 18.0 kg/m2 and 30.0 kg/m2 (inclusive)

   ☞ BMI (body mass index) = {weight (kg) / height (m)2}
3. Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination
4. Subjects considered eligible for the study participation in accordance to the results of vital signs, 12-lead ECG, clinical laboratory tests (including hematology, blood chemistry, urinalysis, serology, etc.) and urine drug screening conducted at the time of screening, based on the investigational product (IP) characteristics (In cases of the results outside the NCS range considered due to irregular lifestyle (drinking, night-time shifts, etc.) final decision of inclusion can be made with additional follow-up after modification of the causal lifestyle)
5. Subjects who has a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period

Exclusion Criteria:

1. Subjects with any clinically significant hepatic, renal, nervous, psychiatric, respiratory, endocrine, circulatory system, neoplastic, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases, or a past medical history of any of the aforementioned conditions.
2. Subjects with a past medical history of gastrointestinal disease (Crohn's disease, ulcers, acute/chronic pancreatitis, etc.) or gastrointestinal surgeries (except for simple appendectomy and hernia repair) which may affect the absorption of the IP.
3. Subjects with clinically significant 12-lead ECG findings including the following results at the time of screening.

   * QTc > 450 ms
   * PR interval > 200 ms
   * QRS duration > 120 ms
4. Subjects with SBP ≥ 150 mmHg or ≤ 90 mmHg; DBP ≥ 100 mmHg or ≤ 60 mmHg; PR ≤ 40 beat/min or ≥ 100 beat/min, when measured in a seated position without an abrupt change in body position for at least 3 minutes.
5. Subjects with laboratory test results as follows.

   * Liver function test (AST, ALT, ALP, γ-GTP and total bilirubin) values exceeding twice the upper limit of normal.
   * Creatinine values outside the reference ranges or eGFR < 60 mL/min/1.73m2
6. Subjects who have participated and given any other study drugs in other clinical study or bioequivalence study within 6 months prior to the first IP administration (the last day of IP administration is considered the end-of-study).
7. Subjects with a past history of drug abuse or a positive urine drug screening test.
8. Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals, within 1 month prior to the first IP administration.
9. Subjects who have taken any prescribed medications or herbal medicine within 2 weeks or any over-the-counter medications or vitamin supplements within 10 days prior to the first IP administration (except for circumstances considered acceptable with no concerned effect on the pharmacokinetics of the IP at the investigator's discretion).
10. Subjects with hypersensitivity reactions or a clinically significant medical history of hypersensitivity reactions to drug substances and additives or other drugs (such as aspirin, anti-biotics, biguanides, etc.).
11. Subjects who have donated whole blood within 2 months or blood components within 1 month or received a blood transfusion within 1 month prior to the first IP administration.
12. Subjects who have consistently drunk alcohol within 6 months exceeding 21 units/week (1 unit= 10 g) prior to the first IP administration or are unable to refrain from drinking from the time of consent until PSV.

    *Alcohol consumption (g) = amount (mL) x alcohol by volume (%) x 0.8* (*pure alcohol 10 g = 12.5 mL)
13. Subjects who have smoked more than 10 cigarettes/day on average 3 months prior to the first IP administration and are unable to oblige the no-smoking rules from 24 hours prior to the first IP administration until the last blood sampling point.
14. Subjects unable to refrain from consuming grapefruit-containing food or beverages from 48 hours prior to the first IP administration until PSV.
15. Subjects unable to refrain from consuming caffeine-containing food or beverages (coffee, green tea, black tea, carbonated drinks, coffee-flavored milk, energy drinks, etc.) from 24 hours prior to the first IP administration until the last blood sampling point.
16. Subjects unable to refrain from vigorous exercise which exceeds daily routine from 48 hours prior to the first IP administration until PSV.
17. Subjects following an unusual diet or unable to consume meals provided during the study.
18. Pregnant subjects with a positive urine HCG test, or lactating female subjects.
19. Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception (administration of contraceptives or transplantation of contraceptives or use of an intrauterine device, infertility surgery (vasectomy or tubule ligation), and physical barriers (spermicide, condom, contraceptive diaphragm, vaginal sponge used with a cervical cap)) from the time of consent until 3months after the last IP administration.
20. Subjects otherwise considered ineligible for participation due to other reasons including clinical laboratory test results not mentioned in the exclusion criteria at the investigator's discretion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Pre-dose (0 hour), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  AUC0-t of ABN401
Cmax | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  Cmax of ABN401

SECONDARY OUTCOMES:
Tmax | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  Tmax of ABN401
AUCinf | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  AUCinf of ABN401
t1/2 | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  t1/2 of ABN401
CL/F | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  CL/F of ABN401
Vd/F | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24h hours (h)post-dose
  Vd/F of ABN401
AUC0-t | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  AUC0-t of ABN401 Metabolite
Cmax | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  Cmax of ABN401 Metabolite
Tmax | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  Tmax of ABN401 Metabolite
AUCinf | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  AUCinf of ABN401 Metabolite
t1/2 | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  t1/2 of ABN401 Metabolite
Metabolic ratio | Pre-dose (0 h), 0.25 hours (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, and 24 hours (h) post-dose
  Metabolic ratio of ABN401

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, Seowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No